CLINICAL TRIAL: NCT04495920
Title: Clinical Evaluation of the Residual Antimicrobial Activity of One Test Product Based on the ASTM E2752 Test Method
Brief Title: Clinical Evaluation of the Residual Antimicrobial Activity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: CAGE Bio Inc. (Industry)
Collaborators: BioScience Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2005367-150
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Bacterial Overgrowth
Keywords: Residual; ASTME2752; Antimicrobial

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Test product (Experimental)
  Interventions: Drug: CGB-S-100

INTERVENTIONS:
Drug: CGB-S-100 — Alcohol and choline geranate
  Other Names: IonLAST gel (CGB-S-100 gel)

SUMMARY:
The purpose of this study is to evaluate the residual antimicrobial efficacy of one test product as defined by the difference between the number of a challenge bacterial species recovered following exposure to the test product and the number recovered when untreated (negative control). The challenge bacterial species to be used is Staphylococcus aureus (ATCC #6538) (S. aureus). Testing will be carried out using a modification of the standardized test method described in ASTM E2752-10 (2015) Standard Guide for Evaluation of Residual Effectiveness of Antibacterial Personal Cleansing Products. Bacterial recoveries will be assayed after application oftest material, using the forearms as a substrate.

DETAILED DESCRIPTION:
At least twelve test subjects (aged 18-65 years), with healthy skin will be used in this study, and will use the test product on one arm, and have the other arm untreated as the negative control. The test sites on both forearms will be inoculated with suspensions containing Staphylococcus au re us (A TCC #653 8), immediately after the 30 minute product drying time, and at approximately 2 hours and 4 hours following test material applications. The test sites will be sampled using the cup scrub procedure approximately 20 minutes following each inoculation. The log 10 microbial recoveries of treated versus untreated sites will be the basis for assessing the residual antimicrobial effectiveness of the test product.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects may be of either sex, between the ages of 18 and 65 years, and of any race.
2. Subjects must possess both forearms.
3. Subjects must have no active skin rashes, dermatoses, or breaks in the skin of the hands or forearms. Subjects must also have no inflammatory skin conditions, such as atopic dermatitis eczema or psoriasis, anywhere on the body
4. Subjects must be in good general health and have no medical diagnosis of a physical condition, such as a current or recent severe illness, a heart murmur, mitral valve prolapse with heart murmur, congenital heart disease, an organ transplant, medicated or uncontrolled diabetes, hepatitis B, hepatitis C, an immunocompromised condition such as AIDS (or HIV positive), lupus, fibromyalgia, ulcerative colitis, Crohn's disease, asthma, heart disease, hypertension, or medicated multiple sclerosis.
5. Subjects must have read and signed an Informed Consent Form, Authorization to Use and Disclose Protected Health Information Form, and List of Restricted Products.

Exclusion Criteria:

1. Participation in a clinical study in the past 7 days or current participation in another clinical study.
2. Experiencing any signs/symptoms of respiratory illness, including cough, fever (body temperature of >100.0 °F) or chills, shortness of breath or difficulty breathing, persistent pain or pressure in the chest, confusion or inability to respond to external stimuli, bluish lips/face, loss of taste/smell, sore throat, headache, nasal discharge ("runny nose"), frequent sneezing, or general fatigue I body aches.
3. Current diagnosis of active Coronavirus Disease 2019 (COVID-19) or have been in close contact within the last 2 weeks of anyone who has been diagnosed as having contracted COVID-19.
4. Travel outside of the state of Montana within the last two weeks.
5. History of smoking or vaping within the last 2 years.
6. Have known allergies or sensitivities to latex (natural rubber), metals, inks, sunscreens, deodorants, laundry detergents, cleansers, soaps, lotions, or common antibacterial agents, particularly, chlorhexidine gluconate (CHG), ethyl alcohol, and isopropyl alcohol or topical antibiotic ointments (e.g., Neosporin® or Polysporin®).
7. Have experienced hives (raised welts) as a reaction to anything that contacted your skin, with the exception of plants known to cause reactions for most humans (e.g., poison oak or poison ivy).
8. Be receiving any topical or systemic antibiotic medications during the 72-hour pre-test conditioning period or on the test day.
9. Be receiving any steroids (including steroid medications used to treat asthma) other than for contraception, hormone therapy, or menopausal purposes during the 72-hour pre-test conditioning period or on the test day.
10. Have any prosthetic joints anywhere in the body or any (pins, screws, plates, rods, or dental implants) anywhere in the body.
11. Have any type of port (or po1iacath) or Peripherally Insetied Central Catheter (PICC).
12. Be nursing a child.
13. Be pregnant, or have plans to become pregnant or impregnate a sexual partner once you have consented to test in this study or during the test period.
14. Any medical condition or use of any medications that, in the opinion of the Principal Investigator, or Consulting Physician should preclude patiicipation.
15. Unwillingness to fulfill the performance requirements of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Significant Log 10 Microbial Change 4 hours post application | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Senior Scientist, Principal Investigator — BIOSCIENCE LAB ORA TORIES, INC.
Locations (1):
- Bioscience Laboratories, Inc., Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No